CLINICAL TRIAL: NCT01215513
Title: An Open-Label, Multi-Centre, Extension Trial, Evaluating the Long-Term Safety and Tolerability of Degarelix One-Month Dosing Regimen in Korean Patients Requiring Androgen Ablation Therapy
Brief Title: Long-Term Safety and Tolerability of Degarelix One-Month Dosing Regimen in Korean Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring Pharmaceuticals Korea, Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS42A
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Degarelix (Experimental)
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix

SUMMARY:
This is an open-label, multi-centre single arm trial to investigate long-term safety and tolerability of degarelix in Korean patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent before any trial-related activity is performed. A trial-related activity is defined as any procedure that would not have been performed during the normal management of the patient
* Has completed the 7-month main trial, FE200486 CS42

Exclusion Criteria:

* Has been withdrawn/discontinued from the FE200486 CS42 trial
* A patient may also not be entered into the CS42A trial at the discretion of the investigator due to safety or lack of efficacy concerns (LH or PSA response) in the CS42 trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (11):
- South Korea (11):
  - Korea University Hospital, Seoul, Anam-dong, Seongbuk-gu
  - Seoul St. Mary's Hospital, Seoul, Banpo-dong, Seocho-gu
  - Kyoungbuk National University Hospital, Daegu, Daegu
  - Yonsei University Health System Gangnam Sevrance, Seoul, Eonguro, Gangnam-gu
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Pyungchon, Gyunggi-do
  - Pusan National University Yangsan Hospital, Mulgeum-eup, Gyungnam
  - Samsung Medical Center, Seoul, Ilwon-dong, Kangnam-gu
  - Asan Medical Center, Seoul, Pungnap-2-dong, Songpa-gu
  - Yonsei University Health System (Sevrance Hospital), Seoul, Seongsanno, Seodaemun-gu
  - Seoul National University Hospital, Seoul, Yeongeon-dong, Chongno-gu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited from 9 sites in Korea. All participants had completed the 7-month main study (CS42, NCT01071915) prior to enrollment into this extension study (CS42A). The CS42A study was conducted between 20 September 2010 (FPFV) and 25 April 2012 (LPLV).
Groups:
- Degarelix: 80 mg degarelix at a concentration of 20 mg/mL were administered as a single 4 mL subcutaneous injection at monthly intervals.
Period: Overall Study
Arm/Group | Degarelix
Started | 157 (157 participants were allocated to treatment in CS42 main study (Intent-to-treat analysis set))
CS42 and CS42A Safety Analysis Set | 156 (156 participants received at least 1 dose of degarelix)
CS42 and CS42A Full Analysis Set | 155 (155 participants received at least 1 dose of degarelix and had at least 1 efficacy assessment)
CS42A Safety Analysis Set | 127 (127 participants were enrolled in the extension study CS42A)
Completed | 112
Not Completed | 45
Not completed — Not completed CS42 | 9
Not completed — Not enrolled from CS42 to CS42A | 21
Not completed — Adverse event (CS42A) | 2
Not completed — Physician decision (CS42A) | 6
Not completed — Withdrawal by subject (CS42A) | 5
Not completed — Miscellaneous reasons (CS42A) | 2

BASELINE CHARACTERISTICS:
Population: The 156 participants included in the CS42 and CS42A saftey analysis set are included in this baseline analysis population.
Arm/Group | Degarelix
Number analyzed (Participants) | 156
Age Continuous [Mean (Standard Deviation); unit: years] | 72.6 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 156
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 156

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Markedly Abnormal Values in Safety Laboratory Variables
Description: The figures present the number of participants who had markedly abnormal levels of safety laboratory variables. Only the laboratory variables that had at least one participant with abnormal value are presented, more variables were included in the study.
  ULN=upper limit of normal
Time Frame: From baseline (day 0) to end of treatment (up to day 364)
Population: Descriptive statistics provided a view of the 1-year safety of degarelix (CS42 and CS42A safety analysis set).
Measure: Number; unit: Participants
Arm/Group | Degarelix
Number analyzed (Participants) | 156
Participants
  S-Alanine aminotransferase (IU/L) >3xULN | 1
  S-Cholesterol (mmol/L) >=8.0 | 1
  S-Potassium (mmol/L) >=5.8 | 10
  S-Sodium (mmol/L) <=130 | 2
  S-Total bilirubin (micromol/L) >1.5xULN | 1
  S-Urea nitrogen (mmol/L) >=10.7 | 10
  B-Basophils (%) >=5 | 1
  B-Eosinophils (%) >=10 | 7
  B-Haematocrit (ratio) <=0.37 | 83
  B-Haemoglobin (g/L) <=115 | 9
  B-Lymphocytes (%) <=10 | 4
  B-Neutrophils (%) >=90 | 1
  B-Red blood cell count (10^12/L) <=3.5 | 25
  B-White blood cell count (10^9/L) <=2.8 | 1
  B-White blood cell count (10^9/L) >=16.0 | 1

2. Primary Outcome: Number of Participants With Markedly Abnormal Values in Vital Signs and Body Weight
Description: This outcome measure included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight. The figures present the number of participants with normal baseline and at least one post-baseline markedly abnormal value.
Time Frame: From baseline (day 0) to end of treatment (up to day 364)
Population: Descriptive statistics provided a view of the 1-year safety of degarelix (CS42 and CS42A safety analysis set).
Measure: Number; unit: Participants
Arm/Group | Degarelix
Number analyzed (Participants) | 156
Participants
  Diastolic blood pressure <=50 and decrease >=15 | 13
  Diastolic blood pressure >=105 and increase >=15 | 0
  Systolic blood pressure <=90 and decrease >=20 | 20
  Systolic blood pressure >=180 and increase >=20 | 1
  Pulse rate <=50 and decrease >=15 | 10
  Pulse rate >=120 and increase >=15 | 0
  Body weight decrease of >=7% from baseline | 4
  Body weight increase of >=7% from baseline | 12

3. Secondary Outcome: Serum Levels of Prostate Specific Antigen (PSA) Over Time
Description: PSA levels were measured over time. The figures present the median level at day 0 (n=155 participants), day 196 (n=148), day 280 (n=115), and day 364 (n=109).
Time Frame: Day 0, day 196, day 280, and day 364
Population: CS42 and CS42A full analysis set (data of all participants who received at least one dose of degarelix and had at least one efficacy assessment after dosing). The figures present the median of the absolute values at day 0 (n=155 participants), day 196 (n=148), day 280 (n=115), and day 364 (n=109).
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Degarelix
Number analyzed (Participants) | 155
ng/mL
  Baseline (Day 0) | 19.2 [1.59 to 100]
  Day 196 | 0.67 [0.1 to 100]
  Day 280 | 0.52 [0.1 to 100]
  Day 364 | 0.46 [0.1 to 100]

4. Primary Outcome: Number of Participants With Markedly Abnormal Values in ECG Variables
Description: This outcome measure included incidence of markedly abnormal changes in ECG variables (PR, QRS, and QT interval, QTcF, and ventricular rate). The figures present the number of participants with normal baseline and at least one post-baseline markedly abnormal value.
Time Frame: From baseline (day 0) to end of treatment (up to day 364)
Population: Descriptive statistics provided a view of the 1-year safety of degarelix (CS42 and CS42A safety analysis set).
Measure: Number; unit: Participants
Arm/Group | Degarelix
Number analyzed (Participants) | 156
Participants
  PR interval (msec) <=120 | 1
  PR interval (msec) >=220 | 3
  QRS interval (msec) >=120 | 3
  QT interval (msec) >=450 | 27
  QT interval (msec) >=480 | 6
  QT interval (msec) >=500 | 2
  QT interval increase of >=30 from baseline | 69
  QT interval increase of >=60 from baseline | 20
  QTcF (msec) >=450 | 25
  QTcF (msec) >=480 | 3
  QTcF (msec) >=500 | 1
  QTcF increase of >=30 from baseline | 39
  QTcF increase of >=60 from baseline | 8
  Ventricular rate (beats/min) <=50 | 1
  Ventricular rate (beats/min) >=120 | 2

ADVERSE EVENTS:
Time Frame: From baseline (day 0) to end of treatment (up to day 364)
Description: The investigator monitored the condition of each participant throughout the study from the time the participant signed the informed consent form until the end of study visit or the end of follow-up period.
Arm/Group | Degarelix
Serious Adverse Events (participants affected / at risk) | 25/156
Other Adverse Events (participants affected / at risk) | 88/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix (N=156)
Angina pectoris (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1)
Hypermetropia (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Metastases to prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Paraplegia (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Removal of internal fixation (Surgical and medical procedures) | 1 (1)
Ureteral stent removal (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix (N=156)
Injection site pain (General disorders) | 39 (55)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 19 (21)
Upper respiratory tract infection (Infections and infestations) | 14 (16)
Constipation (Gastrointestinal disorders) | 13 (13)
Injection site erythema (General disorders) | 13 (13)
Diarrhoea (Gastrointestinal disorders) | 11 (15)
Dizziness (Nervous system disorders) | 11 (13)
Nocturia (Renal and urinary disorders) | 11 (11)
Headache (Nervous system disorders) | 10 (13)
Pollakiuria (Renal and urinary disorders) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10)
Insomnia (Psychiatric disorders) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.